CLINICAL TRIAL: NCT01568749
Title: A Study Investigating the Pharmacokinetic Profiles of Four Extended Release Paracetamol Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: A2750596
Record Dates: First submitted 2011-06-23; First posted 2012-04-02 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-06

CONDITIONS: Analgesia
Keywords: otc; Analgesia; Paracetamol
MeSH Terms: conditions — Agnosia; Ornithine Carbamoyltransferase Deficiency Disease | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Standard paracetamol (Active Comparator): Marketed formulation
  Interventions: Drug: Paracetamol
- Formulation 1 (Experimental): Paracetamol formulation 1
  Interventions: Drug: Paracetamol formulation 1
- Formulation 2 (Experimental): Paracetamol formulation 2
  Interventions: Drug: Paracetamol Formulation 2
- Formulation 3 (Experimental): Paracetamol formulation 3
  Interventions: Drug: Paracetamol formulation 3
- Formulation 4 (Experimental): Paracetamol formulation 4
  Interventions: Drug: Paracetamol formulation 4

INTERVENTIONS:
Drug: Paracetamol — Paracetamol
  Arms: Standard paracetamol
Drug: Paracetamol formulation 1 — Paracetamol
  Arms: Formulation 1
Drug: Paracetamol Formulation 2 — Paracetamol
  Arms: Formulation 2
Drug: Paracetamol formulation 3 — Paracetamol
  Arms: Formulation 3
Drug: Paracetamol formulation 4 — paracetamol
  Arms: Formulation 4

SUMMARY:
A study investigating the pharmacokinetic profiles of four extended release paracetamol formulations

ELIGIBILITY:
Inclusion Criteria:

* Consent:Demonstrates understanding of the study and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.
* Age:Aged 18 to 50 years inclusive.
* Body Mass Index (BMI):Body Mass Index must be in the range 19 - 28 kg/m2.
* Compliance:Understands and is willing, able and likely to comply with all study procedures and restrictions.
* General Health:Good general health with (in the opinion of the investigator) no clinically significant and relevant abnormalities of medical history or physical examination.
* Contraception:Females of childbearing potential who are, in the opinion of the investigator, practicing a reliable method of contraception.

Exclusion Criteria:

* Pregnancy:Women who are pregnant or who have a positive serum pregnancy test.
* Breast-feeding:Women who are breast-feeding.
* Allergy/Intolerance:Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* Clinical Study/Experimental Medication:a) Participation in another clinical study or receipt of an investigational drug within 30 days of the screening visit. b) Previous participation in this study.
* Substance abuse:Recent history (within the last 5 years) of alcohol or other substance abuse.
* Personnel:An employee of the sponsor or the study site or members of their immediate family.
* Disease: a) Current or recurrent disease that could affect the action, absorption or disposition of the study medication or clinical or laboratory assessments (e.g. hepatic disorders, renal insufficiency, congestive heart failure). b) Current or relevant previous history of serious, severe or unstable physical or psychiatric illness, any medical disorder that may require treatment or make the subject unlikely to fully complete the study, or any condition that presents undue risk from the study medication or procedures.
* Vegetarians:Subjects who are vegetarian.
* Hepatitis and HIV Screening:Positive screening for Serum Hepatitis B Surface Antigen, Hepatitis C or Human Immunodeficiency Virus (HIV).
* Medications:Current (within 14 days of screening) or regular use of any prescription, OTC, herbal medicine or drug known to induce or inhibit hepatic drug metabolism in the 30 days prior to dosing, (e.g. barbiturates, theophylline, cimetidine, or erythromycin).
* Smoking:Non-smokers of less than 3 months or current use of nicotine-containing products.
* Blood:Subject has donated or experienced significant blood loss within 56 days of Visit 2, donated plasma within 7 days of Visit 2, or has a hemoglobin value of = 12.0 g/dL.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2008-12; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Disclosure of this information is being delayed to protect business sensitive information. It will be disclosed when it is not longer business sensitive. | Disclosure of this information is being delayed to protect business sensitive information. It will be disclosed when it is not longer business sensitive.

SECONDARY OUTCOMES:
Disclosure of this information is being delayed to protect business sensitive information. It will be disclosed when it is not longer business sensitive. | Disclosure of this information is being delayed to protect business sensitive information. It will be disclosed when it is not longer business sensitive.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- MDS Pharma Services ARIZONA, Phoenix, Arizona, United States